CLINICAL TRIAL: NCT02385370
Title: Bleb Function and Morphology With Intratendon Injection of 0.1 mg MMC in Comparison With Conventional Subtenon Application of 0.02% MMC Soaked Sponges in Trabeculectomy
Brief Title: Bleb Function and Morphology With Intratendon Injection of MMC Compared With Standard Method
Acronym: conj mmc
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Shahid Beheshti Medical University, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92181
Record Dates: First submitted 2015-03-04; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- using standard method of applying MMC (Active Comparator): applying MMC 0.02 % soaked sponges under conjunctival space for 1 to 3 minutes
  Interventions: Drug: MMC
- intratendon injection of MMC (Active Comparator): intratendon injection of 0.1 cc MMC 0.01% at the beginning of the procedure
  Interventions: Drug: MMC

INTERVENTIONS:
Drug: MMC — using 0.02 MMC soaked sponged under the conjunctiva for 1 to 3 minutes
  Arms: using standard method of applying MMC
Drug: MMC — 0.1 cc of 0.01% MMC is injected into the tenon.
  Arms: intratendon injection of MMC

SUMMARY:
Patients with advanced glaucoma that are candidates for trabeculectomy will be included.

Thorough ophthalmic examination including best corrected visual acuity, slit lamp examination, intraocular pressure (IOP) measurement, gonioscopy, funduscopy and specularly microscopy will be performed for all participants. Patients will be assigned randomly to 2 groups. In one group they will undergo fornix based trabeculectomy with conventional MMC 0.02% soaked sponges application. In the other group 0.1 cc of 0.01 MMC will be injected into the tenon at the beginning of the surgery. The rest of the operation is the same for both groups as standard trabeculectomy. Ophthalmic examination including IOP measurement will be performed at one, 3 and 6th month post surgery. Specular microscopy will be requested at final follow up visit. Bleb morphology will be scored according to Indian grading system at 3rd and 6th months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Advanced uncontrolled glaucoma patients.

Exclusion Criteria:

* History of any kind of intraocular surgery.
* Monocular patients.
* Unwillingness to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
IOP (intraocular pressure) | until 6 months
  Goldmann applanation tonometry

SECONDARY OUTCOMES:
Bleb morphology | until 6 months
  scoring the bleb morphologic features according to Indian Grading System

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran, Iran

REFERENCES:
- [Derived] Pakravan M, Esfandiari H, Yazdani S, Douzandeh A, Amouhashemi N, Yaseri M, Pakravan P. Mitomycin C-augmented trabeculectomy: subtenon injection versus soaked sponges: a randomised clinical trial. Br J Ophthalmol. 2017 Sep;101(9):1275-1280. doi: 10.1136/bjophthalmol-2016-309671. Epub 2017 Jan 18. PMID 28100482